CLINICAL TRIAL: NCT01425307
Title: TCD With Transfusions Changing to Hydroxyurea (TWiTCH): A Phase III Randomized Trial to Compare Standard Therapy (Erythrocyte Transfusions) With Alternative Therapy (Hydroxyurea) for the Maintenance of Lowered TCD Velocities in Pediatric Subjects With Sickle Cell Anemia and Abnormal Pre-treatment TCD Velocities
Brief Title: Transcranial Doppler (TCD) With Transfusions Changing to Hydroxyurea
Acronym: TWiTCH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped early due to successfully meeting the primary endpoint
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Boston Children's Hospital (Other); University of Texas Southwestern Medical Center (Other); Children's Healthcare of Atlanta (Other); Children's Hospital of Philadelphia (Other); The Hospital for Sick Children (Other); Children's National Research Institute (Other); Columbia University (Other); St. Jude Children's Research Hospital (Other); University Hospitals Cleveland Medical Center (Other); University of South Alabama (Other); Medical University of South Carolina (Other); University of Alabama at Birmingham (Other); University of Miami (Other); University of Mississippi Medical Center (Other); Wayne State University (Other); Children's Hospital of The King's Daughters (Other); Nemours Children's Clinic (Other); Duke University (Other); East Carolina University (Other); Children's Hospitals and Clinics of Minnesota (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Baylor College of Medicine (Other); State University of New York - Downstate Medical Center (Other); Steven and Alexandra Cohen Children's Medical Center (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-28572 TWiTCH; R01HL095647 (NIH)
Record Dates: First submitted 2011-08-19; First posted 2011-08-30 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2017-05

CONDITIONS: Sickle Cell Anemia
Keywords: Phase III; Sickle cell anemia; Abnormally high Transcranial Doppler velocities.; Reduce risk of primary stroke; Pediatric patients; Chelation therapy
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Therapy (No Intervention): Standard Therapy of monthly transfusions
- Treatment Arm (Experimental): Hydroxyurea will be provided as capsules or liquid
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Capsules (300 mg, 400 mg, or 500 mg) taken once daily liquid formulation (100 mg/mL)
  Other Names: Hydroxycarbamide; Hydrea; Droxia
  Arms: Treatment Arm

SUMMARY:
The primary goal of the Phase III TWiTCH trial is to compare 24 months of alternative therapy (hydroxyurea) to standard therapy (transfusions) for pediatric subjects with sickle cell anemia and abnormally high (≥200 cm/sec) Transcranial Doppler (TCD) velocities, who currently receive chronic transfusions to reduce the risk of primary stroke. For the alternative treatment regimen (hydroxyurea) to be declared non-inferior to the standard treatment regimen (transfusions), after adjusting for baseline differences, the hydroxyurea-treated group must have a mean TCD velocity similar to that observed with transfusion prophylaxis.

DETAILED DESCRIPTION:
Despite the clear results of the STOP and the follow-up STOP II trials, the use of chronic erythrocyte transfusions for primary stroke prevention in children with Sickle Cell Anemia (SCA) remains controversial for many practicing hematologists, as well as for patients and families. Transfusions have proven clinical efficacy in preventing first stroke in children with SCA and abnormal TCD velocities, but their indefinite use may still be difficult to justifY.

The risk of transfusion acquired iron overload is now recognized as a serious consequence of chronic erythrocyte transfusions in children with SCA. After one to two years of monthly transfusions, virtually every patient will have excess hepatic iron deposition that warrants intervention with chelation therapy. The effectiveness of iron chelation has not yet been realized, despite the availability of the oral chelator deferasirox (Exjade®), due to its lack of palatability and increasing recognition of serious drug-related toxicities including renal and hepatic dysfunction. Simply put, indefinite erythrocyte transfusions cannot be viewed as adequate and acceptable long-term therapy for primary stroke prevention in SCA. There is an urgent need to develop an equivalent effective alternative therapy for the prevention of primary stroke in children with SCA, specifically one that better manages iron overload and improves quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric subjects with severe forms of sickle cell anemia (HbSS, HbSβ0 thalassemia,HbSOArab)
2. Age range of 4.0-15.99 years, inclusive, at the time of enrollment
3. Documented index (pre-treatment) abnormally high TCD Velocity by Transcranial Doppler ultrasonography. An abnormally high index TCD is defined as TCD V greater than or equal to 200 cm/sec, or abnormally high TCDi V greater than or equal to185cm/sec, or TCD maximum V greater than or equal to 250 cm/sec.
4. At least 12 months of chronic monthly erythrocyte transfusions since the index abnormal TCD examination
5. Adequate monthly erythrocyte transfusions with average HbS less than or equal to 45% (the upper limit of the established academic community standard) for the past 6 months before enrollment
6. Parent or guardian willing and able to provide informed consent with verbal or written assent from the child
7. Ability to comply with study related treatments, evaluations, and follow-up

Exclusion Criteria:

1. Completed overt clinical stroke or TIA
2. Inability to obtain TCD velocities due to anatomical abnormalities such as a) Inadequate bone windows b) Previous revascularization procedures (e.g., EDAS)
3. Known severe vasculopathy or moya-moya disease on brain MRA
4. Inability to receive or tolerate chronic red blood cell (RBC) transfusion therapy, due to any of the following: a) Multiple RBC alloantibodies making cross-matching difficult or impossible b) RBC autoantibodies making cross-matching difficult or impossible c) Religious objection to transfusions that preclude their chronic use d) Non-compliance with transfusions over the past 6 months before enrollment (temporary exclusion)
5. Inability to take or tolerate daily oral hydroxyurea, including a) Known allergy to hydroxyurea therapy b) Positive serology to HIV infection c) Malignancy d) Current lactation e) Previous stem cell transplant or other myelosuppressive therapy
6. Clinical and laboratory evidence of hypersplenism (temporary exclusions): a) Palpable splenomegaly greater than 5cm below the left costal margin AND b) Transfusion requirement greater than 250 mL/kg over the previous 12 months
7. Abnormal laboratory values at initial evaluation (temporary exclusions): a) Pre-transfusion hemoglobin concentration less than 8.0 gm/dL b) WBC count less than 3.0 x 10^9/L c) Absolute neutrophil count (ANC) less than 1.5 x 10^9/L d) Platelet count less than 100 x 10^9/L e) Serum creatinine more than twice the upper limit for age OR greater than or equal to 1.0 mg/dL
8. Current participation in other therapeutic clinical trials
9. Current use of other therapeutic agents for sickle cell disease (e.g., arginine, decitabine, magnesium). Subjects must have been off hydroxyurea for at least 3- months prior to enrollment.
10. Any condition or chronic illness, such as a positive tuberculin (PPD) test, which in the opinion of the CI makes participation ill-advised.
11. Inability or unwillingness to complete required screening and exit studies, including TCD ultrasonography, brain MRI/MRA, liver MRI and blood tests.
12. A sibling enrolled in TWiTCH
13. Pregnancy or unwillingness to use a medically acceptable form of contraception if sexually active (male OR female).

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2011-08; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell E. Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ware RE, Davis BR, Schultz WH, Brown RC, Aygun B, Sarnaik S, Odame I, Fuh B, George A, Owen W, Luchtman-Jones L, Rogers ZR, Hilliard L, Gauger C, Piccone C, Lee MT, Kwiatkowski JL, Jackson S, Miller ST, Roberts C, Heeney MM, Kalfa TA, Nelson S, Imran H, Nottage K, Alvarez O, Rhodes M, Thompson AA, Rothman JA, Helton KJ, Roberts D, Coleman J, Bonner MJ, Kutlar A, Patel N, Wood J, Piller L, Wei P, Luden J, Mortier NA, Stuber SE, Luban NLC, Cohen AR, Pressel S, Adams RJ. Hydroxycarbamide versus chronic transfusion for maintenance of transcranial doppler flow velocities in children with sickle cell anaemia-TCD With Transfusions Changing to Hydroxyurea (TWiTCH): a multicentre, open-label, phase 3, non-inferiority trial. Lancet. 2016 Feb 13;387(10019):661-670. doi: 10.1016/S0140-6736(15)01041-7. Epub 2015 Dec 6. PMID 26670617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 3 First Patient In: 16-Sep-2011; Last Patient Last Visit 10-Feb-2015
  26 medical institutions in the United States of America and Canada
Pre-assignment Details: 159 were enrolled. 121 met eligibility criteria and randomized to treatment.
Groups:
- Treatment Arm: Hydroxyurea will be provided as capsules or liquid
  Hydroxyurea: Capsules (300 mg, 400 mg, or 500 mg) taken once daily or liquid formulation (100 mg/mL)
Period: Overall Study
Arm/Group | Standard Therapy | Treatment Arm
Started | 61 (Randomized Sample: 61; Intention-to Treat Sample:61) | 60 (Randomized Sample: 60; Intention-to Treat Sample:60)
Completed | 42 (Treatment Phase: 42; 6-Month Follow up: 58) | 41 (Treatment Phase: 41; 6-Month Follow-up:59)
Not Completed | 19 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy | Treatment Arm | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 61 | 60 | 121
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (2.6) | 9.7 (3.2) | 9.6 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 29 | 71
  Male | 19 | 31 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 58 | 57 | 115
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 58 | 57 | 115
  White | 0 | 1 | 1
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 5 | 9
  United States | 57 | 55 | 112
Age at Index TCD [Mean (Standard Deviation); unit: years] — The index TCD is the documented first abnormal TCD examination. This TCD examination was at least 12 months prior to eligibility for TWiTCH.
  years | 5.7 (2.0) | 5.0 (1.8) | 5.4 (1.9)
Duration of Transfusions [Mean (Standard Deviation); unit: years] — Duration of Transfusions refers to the duration of chronic transfusion therapy (either simple, partial exchange or erythrocytapheresis) for primary stroke prevention.
  years | 3.8 (1.8) | 4.5 (2.8) | 4.1 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Difference in TCD Time-averaged Mean Velocity (TAMV) on the Index Side
Description: The primary endpoint for the TWiTCH trial was the difference between the treatment groups of the maximum TCD TAMV on the index side, calculated from a mixed model. The index side is the side with the higher mean (averaged over baseline evaluations) of the maximum (over arteries on that side) TCD time-averaged velocity. Values of the TAMV on the index site were obtained at clinic visits during baseline and during the treatment period.
Time Frame: Since the study was terminated early, time frame is from beginning of treatment until end of treatment (up to 24 Months).
Population: Intention-to-Treat
Measure: Mean (95% Confidence Interval); unit: cm/sec
Arm/Group | Treatment Arm | Standard Therapy
Number analyzed (Participants) | 60 | 61
cm/sec | 138 [135 to 142] | 143 [140 to 146]
Statistical Analysis 1: Comparison: Treatment Arm vs Standard Therapy; Participants were randomized at a central site, stratified by site with a block size of four, and an adaptive randomization scheme was used to balance the covariates of baseline age and TCD velocity. The treatment period lasted 24 months. The primary study endpoint was the 24 month TCD velocity calculated from a general linear mixed model, with the non-inferiority margin set at 15 cm/s. The primary analysis was done in the intention-to-treat population; Test type: Non-Inferiority or Equivalence — We hypothesized that the Alternative arm mean TCD velocity at 24 months will be less than the Standard arm mean TCD velocity plus 15cm/sec. We used Lan-DeMets boundaries to control overall Type I error rate at α = 0.05. For looks at exactly 1/3, 2/3, and 100 percent of the completed subjects, the cumulative α were estimated to be 0.0001, 0.001, and 0.05, respectively; p < 0.05, Mixed Models Analysis — P value for non inferiority was 8.82 X 10^-16; Linear mixed model; Mean Difference (Final Values) = 4.54, 95% CI 2-sided [0.10 to 8.98]

2. Secondary Outcome: TCD Time-averaged Mean Velocity on the Non-index Side
Description: This secondary endpoint for the TWiTCH trial will be maximum TCD time-averaged mean velocity on the non-index side. The non-index side is the side with the lower mean (averaged over baseline evaluations) of the maximum (over arteries on that side) TCD time-averaged velocity. Values of the secondary endpoint will be obtained at clinic visits during baseline and during the 24-month treatment period.
Time Frame: 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Primary Stroke Events
Description: This secondary outcome measure will compare standard to alternative therapy for primary stroke events (a) primary ischemic stroke; b) primary hemorrhagic stroke
Time Frame: 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Non-stroke Neurological Events
Description: This secondary objective will compare standard to alternative treatment for the incidence of non-stroke neurological events. Data for this outcome will be collected through entry and exit neurological exams.
Time Frame: 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Change of Baseline in Hepatic Iron Overload as Assessed by Serum Ferritin
Description: This secondary objective will compare standard to alternative therapy for hepatic iron overload.
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: ng per mL
Groups:
- Treatment Arm: Hydroxyurea will be provided as capsules and liquid
Arm/Group | Standard Therapy | Treatment Arm
Number analyzed (Participants) | 61 | 60
ng per mL | -38 (2095) | -1805 (1651)
Statistical Analysis 1: Comparison: Standard Therapy vs Treatment Arm; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Effects on Quality of Life
Description: Standard Quality of Life measure will be taken during specific time points as well as one newly developed Sickle Cell Disease-specific test.
Time Frame: 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Functional Status
Description: This outcome will be measured using Barthel Index testing at the beginning, middle, and end of the treatment period.
Time Frame: 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Neuropsychological Decline
Description: This outcome will be measured using standardized neurocognitive tests at baseline and exit.
Time Frame: 24 months
Reporting Status: Not Posted

9. Secondary Outcome: Growth and Development
Description: This outcome will be measured by capturing height and weight monthly and conducting an annual pubertal assessment.
Time Frame: 24 months
Reporting Status: Not Posted

10. Secondary Outcome: Number of Participants With Transfusion Events
Description: This outcome will be recorded on every interval visit form through questions asking whether there have been transfusion complications. Any complication higher than a CTCAE grade 2 event will be reported as a SAE.
Time Frame: 24 months
Reporting Status: Not Posted

11. Secondary Outcome: Number of Participants With Hydroxyurea Toxicities
Description: This measure will be performed on a monthly basis throughout the trial by recording the CBC and retic count.
Time Frame: 24 Months
Reporting Status: Not Posted

12. Secondary Outcome: Number of Participants With Phlebotomy Complications
Description: This outcome will be recorded on every interval visit form through questions asking whether there have been phlebotomy complications. Any complication higher than a CTCAE grade 2 event will be reported as a SAE.
Time Frame: 24 months
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants With Liver MRI Complications
Description: This outcome will be recorded through questions asking whether there have been Liver MRI complications at baseline, middle, and end of treatment. Any complication higher than a CTCAE grade 2 event will be reported as a SAE.
Time Frame: 24 months
Reporting Status: Not Posted

14. Secondary Outcome: Number of Participants With Serious Adverse Events
Time Frame: 24 Months
Reporting Status: Not Posted

15. Secondary Outcome: Change of Baseline in Hepatic Iron Overload as Assessed by Liver Iron Concentration
Description: This secondary objective will compare standard to alternative therapy for hepatic iron overload.
Time Frame: Baseline and 24 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: mg FE per g dry weight liver
Arm/Group | Standard Therapy | Treatment Arm
Number analyzed (Participants) | 52 | 58
mg FE per g dry weight liver | 2.4 (8.7) | -1.9 (4.2)
Statistical Analysis 1: Comparison: Standard Therapy vs Treatment Arm; Test type: Superiority or Other; p = 0.0011, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Standard Therapy | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 6/61 | 9/60
Other Adverse Events (participants affected / at risk) | 53/61 | 58/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=61) | Treatment Arm (N=60)
Vaso-occlusive Pain (Blood and lymphatic system disorders) | 1 (3) | 5 (11)
Fever (Infections and infestations) | 1 (1) | 4 (4)
Acute Chest Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (5)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Intracranial Aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Splenomeagaly/Splenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=61) | Treatment Arm (N=60)
Sickle Cell Anemia with Crisis (Blood and lymphatic system disorders) | 9 (28) | 24 (62)
Abdominal Pain (Gastrointestinal disorders) | 7 (12) | 6 (7)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 3 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (6)
Gastritis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (7)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pyrxia (General disorders) | 7 (7) | 10 (10)
Seasonal Allergy (Immune system disorders) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Gastrointestinal Viral Infection (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 3 (4) | 7 (9)
Pharyngitis (Infections and infestations) | 0 (0) | 5 (5)
Pharyngitis Streptococcal (Infections and infestations) | 9 (12) | 9 (11)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 14 (21) | 18 (30)
Urinary Tract Infection (Infections and infestations) | 6 (6) | 3 (4)
Viral Infection (Infections and infestations) | 10 (11) | 9 (12)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 3 (3)
Procedural Dizziness (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Transfusion Reaction (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Alanine Aminotranferase (Investigations) | 12 (16) | 7 (11)
Aspartate Aminotranserase (Investigations) | 9 (11) | 14 (16)
Blood Bilirubin Increased (Investigations) | 12 (37) | 3 (4)
Blood Creatinine Increased (Investigations) | 0 (0) | 7 (8)
Coombs Direct Test Positive (Investigations) | 7 (10) | 3 (4)
Hemoglobin Decreased (Investigations) | 25 (66) | 32 (76)
Neutrophil Count Decreased (Investigations) | 0 (0) | 15 (19)
Platelet Count Decreased (Investigations) | 0 (0) | 4 (4)
Reticulocyte Count Decreased (Investigations) | 0 (0) | 12 (16)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Headache (Nervous system disorders) | 19 (38) | 22 (41)
Migraine (Nervous system disorders) | 3 (3) | 7 (9)
Acute Chest Syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Poor Venous Access (Vascular disorders) | 4 (4) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
Further analysis is required to verify that the Adverse Events are accurately represented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less